CLINICAL TRIAL: NCT05309928
Title: A Rational Approach to the Identification of New Treatment Options to Prevent Congenital Syphilis: Phase 1 Study of the Pharmacokinetics of Amoxicillin in Pregnancy
Brief Title: Phase 1 Study of the Pharmacokinetics of Amoxicillin in Pregnancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jodie A. Dionne, MD, Associate Professor of Medicine; Division of Infectious Diseases, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-300008691; UAB (Other: UAB)
Record Dates: First submitted 2022-03-14; First posted 2022-04-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Related
Keywords: pharmacokinetics; amoxicillin
MeSH Terms: interventions — Amoxicillin; Probenecid

STUDY DESIGN:
Intervention Model Description: The study design is a prospective phase I pharmacokinetic study focused on dosing of 500 mg oral amoxicillin administration in pregnant women in the 2nd and 3rd trimester.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Amox 500 mg (Experimental): Amoxicillin 500 mg PO
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — medication administration
  Other Names: Probenecid

SUMMARY:
The study design is a prospective phase I pharmacokinetic study focused on dosing of 500 mg oral amoxicillin administration in pregnant women in the 2nd and 3rd trimester.

DETAILED DESCRIPTION:
Twenty adult pregnant women in good health who are admitted for preterm premature rupture of membranes (24-34 weeks gestational age) will be enrolled in this intensive pharmacokinetic study. Basic information will be collected from the medical record including age, weight, height, pregnancy dating, medications, and allergies.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant, engaged in prenatal care with a medical provider (at least one visit)
2. Estimated gestational age 24-34 weeks
3. Able to provide informed consent
4. English speaking

Exclusion Criteria:

1. Receipt of amoxicillin within the past 7 days. (Routine GBS prophylaxis with ampicillin or other antibiotic and routine surgical prophylaxis prior to cesarean with cephalexin and azithromycin 500 mg IV is allowed).
2. Known hypersensitivity or intolerance of amoxicillin, penicillin, other beta lactam or cephalosporin antibiotics.
3. Known renal impairment (serum creatinine ≥1.2 mg/dL).
4. Active concomitant medications known to interact with amoxicillin: allopurinol, methotrexate, mycophenolate, immune checkpoint inhibitors (ie. pembrolizumab), tetracyclines (ie. doxycycline), vitamin K antagonists (ie. warfarin), aminoglycosides (ie. gentamicin).

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change of Amoxicillin Level in Plasma during Pregnancy | 0, 1, 2, 3, 4, 6, 8 hours after medication administration
  quantitative drug level in blood
Amoxicillin Level in Cord Blood | at delivery
  quantitative drug level in cord blood to calculate transplacental transfer rate for amoxicillin
Change of Amoxicillin Level in Plasma in the Postpartum state | 0, 1, 2, 3, 4, 6, 8 hours after medication administration
  quantitative drug levels in blood to compare to pregnancy state values

SECONDARY OUTCOMES:
additional pharmacologic measures | 1-8 hours after administration
  1. Maximum concentration (Cmax) in maternal serum.
Additional pharmacologic measure | 1-8 hours after administration
  time to maximum concentration (tmax) in maternal serum

CONTACTS AND LOCATIONS:
Overall Officials: Jodie Dionne, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States